CLINICAL TRIAL: NCT02628730
Title: Pulmonary Vein Reconnection Following Ablation Index-guided Ablation: a Success Evaluation (PRAISE)
Brief Title: Pulmonary Vein Reconnection Following Ablation Index-guided Ablation: a Success Evaluation
Acronym: PRAISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWI-IIS-386; NHS REC (Registry Identifier: 193216/878714/1/459)
Record Dates: First submitted 2015-11-20; First posted 2015-12-11 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ablation; Pulmonary vein isolation; Ablation Index
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation Index Group (Active Comparator): PVI using radiofrequency ablation (RFA) guided by Ablation Index.
  Interventions: Device: PVI using ThermoCool® SmartTouch® Catheter
- Reference Group (Contact Force Group) (Other): That group will be formed by the 40 patients who underwent mandatory repeat EPS 8-10 weeks following contact force guided PVI in the PRESSURE study (ClinicalTrials.gov Identifier: NCT01942408). RFA ablation data from reference group (Contact Force Group) will be compared with those obtained from the Ablation Index Group.
  Interventions: Device: RFA ablation data comparison

INTERVENTIONS:
Device: PVI using ThermoCool® SmartTouch® Catheter — PVI using RFA, using ThermoCool® SmartTouch® Catheter (Biosense Webster Inc., CA, US), guided by Ablation Index.
  Arms: Ablation Index Group
Device: RFA ablation data comparison — Ablation data from previous ablations, using ThermoCool® SmartTouch® Catheter (Biosense Webster Inc., CA, US), that members of this group had in the past, will be compared with those of the Active Comparator Group.
  Arms: Reference Group (Contact Force Group)

SUMMARY:
Atrial fibrillation (AF) is the commonest condition affecting the rhythm of the heart. Tablets to try to normalise the heart rhythm rarely work well. As a result, doctors have devised a treatment called catheter ablation in which special wires are used to deliver heat energy (called ablation lesions) on the inside surface of the heart. Unfortunately, in many patients (almost 1 in 2), some of these ablation lesions recover, and this leads to AF recurrence. Many of these patients then need a second procedure to deliver further ablation at these recovered areas.

Recent research has shown that monitoring of heat delivery with a factor called Ablation Index may be useful in predicting which ablation lesions are less likely to recover. Therefore, we aim to carry out AF ablation guided with Ablation Index (AI) and observe whether this will be associated with better durability of ablation lesions, and thereby better freedom from AF.

This study will include patients with persistent AF, those whose AF episode(s) last for longer than seven days. All patients participating in the study will undergo an initial ablation treatment guided by ablation Index . All patients will undergo a repeat procedure 8-10 weeks after their initial treatment. Any gaps found during the second procedure will be closed again by delivery of ablation.

All participants will be issued with a simple to use handheld heart rhythm monitor, and asked to make a 30-second recording of their heart rhythm each day and also whenever they have symptoms. The monitor stores these recordings and they will be downloaded at review appointments arranged 6 weeks, 3 months, 6 months and 12 months after the initial ablation procedure.

DETAILED DESCRIPTION:
The study is a prospective cohort study in 40 patients with Persistent AF. It will comprise two groups:

1. Active Group (AI guided ablation): An initial pulmonary vein isolation (PVI) procedure will be performed guided by AI targets. All patients (regardless of AF recurrence) will undergo a repeat EP study at 8-10 weeks to identify and re-ablate site(s) of PV reconnection
2. Historical control group (Contact Force Guided Ablation): will be formed by the 40 patients enrolled to the repeat study arm of the PRESSURE study (ClinicalTrials.gov Identifier: NCT01942408). All 40 patients underwent contact force-guided PVI followed by a repeat EP study after 8-10 weeks.

End-points

Primary outcome measure:

The proportion of patients with pulmonary vein (PV) reconnection seen at repeat EP study

Secondary outcome measures:

* The proportion of reconnected PVs seen at repeat electrophysiology (EP) study
* The proportion of patients maintaining freedom from atrial tachyarrhythmia for 12 months (after an initial 12 week blanking period)
* QOL 6 and 12 months after initial ablation, as quantified by the validated atrial Fibrillation Effect on QualiTy-of-life (AFEQT) and EQ-5D-5Lquestionnaires.
* Rates of major complications occurring within 60 days after a PVI procedure, measured in composite numbers and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Persistent AF (defined, according to the ESC/EHRA Guidelines for the Management of Atrial Fibrillation 2010, as AF episode that either lasts longer than 7 days or requires termination by cardioversion, either with drugs or by direct current cardioversion (DCC) ).
* Symptomatic in spite of drug treatment
* Due to undergo pulmonary vein isolation by RF ablation

Exclusion Criteria:

* Inability or unwillingness to receive oral anticoagulation with a Vitamin K antagonist (VKA) or non-VKA (NOAC) agent
* Previous catheter or surgical ablation procedure for AF
* Unwillingness or inability to complete the required follow-up arrangements
* Current pattern of paroxysmal AF
* Long standing persistent AF (continuous AF longer than 12 months before ablation)
* Prior prosthetic mitral valve replacement or severe structural cardiac abnormality
* Known infiltrative cardiomyopathy
* Known severe left ventricular systolic function (ejection fraction <35%)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with PV reconnection seen at repeat EP study | 8-10 weeks

SECONDARY OUTCOMES:
The proportion of reconnected PVs seen at repeat EP study | 8-10 weeks
The proportion of patients maintaining freedom from atrial fibrillation. | 12 months
Quality of Life (QOL) using score of AFEQT Questionnaire. | 6 and 12 months
  AFEQT score will be obtained as the sum of units on the questionnaire's scale.
QOL using score of EQ-5D-5L Questionnaire. | 6 and 12 months
  EQ-5D-5L score will be obtained as the sum of units on the questionnaire's scale.
Major complications percent. | Occurring within 60 days after a PVI procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MD, DM, FRCP, Study Chair — Liverpool Heart and Chest Hospital, Liverpool, UK; Ahmed A Hussein, MRCP, MSc, Principal Investigator — Liverpool Heart and Chest Hospital, Liverpool, UK; Moloy Das, Principal Investigator — Freeman Hospital, Newcastle, UK; Antonio D Russo, Principal Investigator — Centro Cardiologico Monzino
Locations (3):
- Centro Cardiologico Monzino, IRCCS,, Milan, Italy
- United Kingdom (2):
  - Liverpool Heart & Chest Hospital NHS Foundation Trust, Liverpool
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Background] Das M, Wynn GJ, Morgan M, Lodge B, Waktare JE, Todd DM, Hall MC, Snowdon RL, Modi S, Gupta D. Recurrence of atrial tachyarrhythmia during the second month of the blanking period is associated with more extensive pulmonary vein reconnection at repeat electrophysiology study. Circ Arrhythm Electrophysiol. 2015 Aug;8(4):846-52. doi: 10.1161/CIRCEP.115.003095. Epub 2015 Jun 24. PMID 26108982
- [Derived] Hussein A, Das M, Riva S, Morgan M, Ronayne C, Sahni A, Shaw M, Todd D, Hall M, Modi S, Natale A, Dello Russo A, Snowdon R, Gupta D. Use of Ablation Index-Guided Ablation Results in High Rates of Durable Pulmonary Vein Isolation and Freedom From Arrhythmia in Persistent Atrial Fibrillation Patients: The PRAISE Study Results. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006576. doi: 10.1161/CIRCEP.118.006576. PMID 30354288
- See also: The Effect of Early Repeat Atrial Fibrillation (AF) Ablation on AF Recurrence (PRESSURE) Study — https://clinicaltrials.gov/ct2/show/NCT01942408?term=Dhiraj&rank=2